CLINICAL TRIAL: NCT03061513
Title: Ubiquinol in Parkinson's Disease: Safety, Tolerability, and Effects Upon Oxidative Damage and Mitochondrial Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1112012060
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; ubiquinol; CoQ10; magnetic resonance spectroscopy; lactate; glutathione
MeSH Terms: conditions — Parkinson Disease | interventions — ubiquinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ubiquinol (Active Comparator): 600mg ubiquinol daily for 24 weeks
  Interventions: Drug: Ubiquinol
- Placebo (Placebo Comparator): Placebo daily for 24 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Ubiquinol — Ubiquinol caplets 600mg/day
  Arms: Ubiquinol
Dietary Supplement: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether ubiquinol is well tolerated, can affect the symptoms of Parkinson's Disease and change the energy levels in the brain. Subjects will be randomized to taking ubiquinol or placebo and will have a neurological evaluation, magnetic resonance spectroscopy (MRS) and blood test for biological markers taken during the study.

DETAILED DESCRIPTION:
Multiple lines of evidence have implicated abnormal energy metabolism and deficient mitochondrial function in Parkinson's disease, presenting a unique target for therapy. A pilot study of ubiquinol in PD was therefore undertaken to determine its effects upon physiologic measures of mitochondrial metabolic function. The incorporation of a neuroimaging biomarker is particularly important, since changes would demonstrate our ability to achieve Central Nervous System (CNS) access from this an formulation, accompanied by a meaningful neurophysiologic effect. Hydrogen Proton Magnetic Resonance Spectroscopy Imaging (1H MRSI) is a technique that provides insight into the metabolism of several endogenous brain compounds, most notably N-acetyl-L-aspartate (NAA), choline-containing compounds (Cho), and creatine and phosphocreatine (Cr). A number of studies of mitochondrial function have now firmly established the utility of 1H MRSI in probing potential mitochondrial energy metabolism dysfunction, in primary mitochondrial disorders, but also in PD. This pilot study is therefore designed to test whether oral ubiquinol affects cerebral indices of mitochondrial dysfunction, as measured by 1H MRSI in patients with Parkinson's disease, and to gather preliminary information on the safety and tolerability of ubiquinol in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PD according to the Untied Kingdom (UK) Brain Bank Criteria, and confirmed by a Movement Disorders neurologist;
* age 40-75 years; diagnosis within 5 years of study participation;
* PD medications able to remain at stable doses in the opinion of the enrolling investigator;
* able to undergo MRI;
* absence of significant medical, psychiatric, and other neurological disease;
* absence of dementia and Mini-Mental State Examination (MMSE) > 26.

Exclusion Criteria:

* failure to meet diagnosis by above criteria;
* time since diagnosis > 5 years before study participation;
* PD medications not predicted to remain at stable doses in the opinion of the enrolling investigator;
* unable to undergo MRI;
* unable to comply with informed consent process;
* presence of significant medical, psychiatric (including major depressive disorder) or other neurological (including epilepsy, brain tumor, stroke) disease;
* diagnosis of dementia and/or MMSE 26 or lower;
* possibility of pregnancy (negative test required in women of childbearing age);
* taking medications including antipsychotic agents and dopamine- blocking anti-emetic agents;
* taking Coenzyme Q10;
* participation in another clinical trial within the last 3 months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Henchcliffe, MD DPhil, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from the clinical practice at Weill Cornell Medicine's (WCM) Parkinson's Disease Department as well as Weill Cornell Medicine, and utilized flyers.
Pre-assignment Details: One screening visit consisting of: neurological examination, interview on health topics, and questionnaires on health topics.
Period: Overall Study
Arm/Group | Ubiquinol | Placebo
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ubiquinol | Placebo | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 2 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: The incidence and severity of adverse events in Parkinson disease patients taking 600mg ubiquinol or placebo daily over a 6 month period.
Time Frame: at 24 weeks
Population: ITT
Measure: Number; unit: Number of Adverse Events
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 6 | 5
Number of Adverse Events | 27 | 12

2. Secondary Outcome: Cerebral Redox Markers
Description: Change from baseline in lactate levels at 8 weeks as determined by Magnetic Resonance Spectroscopy
Time Frame: at baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Ubiquinol | Placebo
Number analyzed (Participants) | 6 | 4
Ratio | -11.98 (18.57) | 6.23 (23.19)

ADVERSE EVENTS:
Arm/Group | Ubiquinol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 5/6 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ubiquinol (N=6) | Placebo (N=5)
Fever (General disorders) | 0 | 1
Motor Vehicle Accident (General disorders) | 0 | 1
Common Cold Syndrome (Infections and infestations) | 3 | 2
Dizziness (General disorders) | 4 | 0
Sleepiness (General disorders) | 4 | 1
Skin rash, itching (Skin and subcutaneous tissue disorders) | 1 | 1
Nausea (General disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Upset stomach (Gastrointestinal disorders) | 0 | 1
Cognitive decline (Nervous system disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Moodiness (General disorders) | 1 | 0
Stomatitis (General disorders) | 0 | 1
Lumbar pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Sudden falls (General disorders) | 1 | 0
Peripheral edema (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No